CLINICAL TRIAL: NCT06910644
Title: Dexmedetomidine Versus Lidocaine Infusions as Adjuvants to General Anesthesia for Chronic Pain Management After Mastectomy: A Randomized Controlled Trial
Brief Title: Dexmedetomidine Versus Lidocaine Infusions as Adjuvants to General Anesthesia for Chronic Pain Management After Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsaid Abdel Fattah, Lecturer of Anesthesia, Surgical ICU and Pain Management, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2411-501-087-193
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Dexmedetomidine; Lidocaine; Infusion; Adjuvants; General Anesthesia; Chronic Pain; Mastectomy
MeSH Terms: conditions — Chronic Pain | interventions — Dexmedetomidine; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group (Experimental): Patients will receive 1 μg/kg of intravenous dexmedetomidine over 10 min followed by an intravenous infusion of 0.5 μg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Lidocaine group (Experimental): Patients will receive a bolus of intravenous lidocaine 1.5mg/kg over 10 min followed by a continuous infusion of lidocaine 1.5mg/kg/h.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Patients will receive intravenous isotonic saline 0.9% in the same volume and manner as the study drugs.
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive 1 μg/kg of intravenous dexmedetomidine over 10 min followed by an intravenous infusion of 0.5 μg/kg/h.
  Arms: Dexmedetomidine group
Drug: Lidocaine — Patients will receive a bolus of intravenous lidocaine 1.5mg/kg over 10 min followed by a continuous infusion of lidocaine 1.5mg/kg/h.
  Arms: Lidocaine group
Drug: Isotonic saline — Patients will receive intravenous isotonic saline 0.9% in the same volume and manner as the study drugs.
  Arms: Control group

SUMMARY:
This study aims to compare dexmedetomidine and lidocaine infusions as adjuvants to general anesthesia for chronic pain management after mastectomy.

DETAILED DESCRIPTION:
Chronic pain after breast cancer surgery is a significant problem that is expected to become more relevant because the number of patients undergoing breast cancer surgery is increasing owing to the longer survival associated with this surgery.

Lidocaine is the local anesthetic, which is used more often, and it is considered the prototype of amino-amide local anesthetics. Dexmedetomidine (DEX) is a highly selective agonist that acts by binding with presynaptic alpha 2-adrenergic receptor and then activating the negative feedback loop of the sympathetic nerve response, leading to inhibited norepinephrine release from the sympathetic terminals and decreased reflex activity of the sympathetic nervous.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years.
* American Society of Anesthesiologists (ASA) physical status II.
* Scheduled for mastectomy with axillary dissection (either modified radical mastectomy with or without latissimus dorsi flap or conservative breast surgery) due to breast cancer.

Exclusion Criteria:

* Patient refusal.
* Known allergy to any of the study drugs.
* Those with hepatic or renal insufficiency.
* Patients who are running regularly on B blockers.
* α2 adrenergic agonists and sedatives.
* Psychoactive medications.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women scheduled for mastectomy
Enrollment: 90 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the chronic pain | 6 months postoperatively
  Incidence of the chronic pain will be recorded.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 48 hours postoperatively
  Time to the 1st rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Heart rate | Till the end of operation (Up to 2 hours)
  Heart rate will be recorded before infusion (Baseline value), 5,10, 15, 30, 45 and 60 minutes and at the end of operation.
Mean arterial pressure | Till the end of operation (Up to 2 hours)
  Mean arterial pressure will be recorded before infusion (Baseline value), 5,10, 15, 30, 45 and 60 minutes and at the end of operation.
Total morphine consumption | 48 hours postoperatively
  Rescue analgesia of morphine 0.1 mg/kg/dose (max 0.3 mg/kg/day) boluses will be given if the visual analogue scale (VAS)>3.
Degree of pain | 12 weeks postoperatively
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at PACU, 1, 2, 4, 6, 8, 12, 18, 24, 36, 48 h,1, 2, 3, 4, 8, and 12 weeks postoperatively.
Incidence of post-mastectomy pain syndrome | 6 months postoperatively
  Incidence of post-mastectomy pain syndrome will be recorded.
Activity level | 12 weeks postoperatively
  The activity level will be assessed using the Barthel Activities of Daily Living scale (ADL) 2, 3, 4, 8 and 12 weeks postoperatively. This scale comprises 10 basic daily activities (bowel, bladder, feeding, toilet, bathing, dressing, grooming, walking, stairs and transfer) with each item scored as 0 = need complete help, 1 = need some help or 2 = need no help .
Assessment of quality of life | 12 weeks postoperatively
  Quality of life will be assessed using the Flanagan Quality of Life Scale (QOLS), which is a 16-item (domain) questionnaire with each item scored from 1 to 7 points. The scale will be explained to the patients by the pain physician, and the total score will be calculated and recorded at the preoperative assessment (baseline) and at 2, 3, 4, 8 and 12 weeks postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.